CLINICAL TRIAL: NCT01183650
Title: A Study to Evaluate the Pharmacokinetics of Tadalafil Administered Once Daily in Japanese and Non-Japanese Subjects With Benign Prostatic Hyperplasia
Brief Title: A Study of Tadalafil in Benign Prostatic Hyperplasia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 13910; H6D-MC-LVIY (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-08-13; First posted 2010-08-17 (Estimated); Results first posted 2012-05-16 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-04

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tadalafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tadalafil (Experimental): 5 mg, administered orally, daily for 10 days
  Interventions: Drug: Tadalafil

INTERVENTIONS:
Drug: Tadalafil — 5 mg, administered orally, daily for 10 days
  Other Names: LY450190; Cialis; Adcirca

SUMMARY:
The purpose of this study is to investigate the pharmacokinetics of tadalafil in Japanese and non-Japanese men with Benign Prostatic Hyperplasia (BPH).

The safety of tadalafil will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Have had lower urinary tract symptoms secondary to benign prostatic hyperplasia (BPH-LUTS) (as diagnosed by a qualified physician) >6 months at screening visit. Lower urinary tract symptoms (LUTS) include those associated with voiding (obstructive symptoms, such as incomplete emptying, intermittency, weak stream, straining) and/or storage (irritative symptoms, such as frequency, urgency, nocturia).
* Have BPH-LUTS with moderate-to-severe symptoms confirmed by an International Prostate Symptom Score (IPSS) >12. (The IPSS total score is defined as the sum of Questions 1 through 7 and does not include the IPSS Quality of Life.)
* Taking into account the age and disease status, subjects determined to be in good health according to medical history, physical examination, electrocardiogram (ECG), and laboratory safety assessments.
* Body mass index between 18 and 30 kg/m^2 inclusive.
* Agree not to use any other approved or experimental pharmacologic BPH, erectile dysfunction (ED), and/or overactive bladder (OAB) treatments, including alpha blockers, phosphodiesterase type 5 (PDE5) inhibitors, or herbal preparations at least 1 week prior to dosing and through to follow-up.
* Subjects with a serum prostate-specific antigen (PSA) <10.0 ng/mL. Subjects with a serum PSA greater than or equal to 4.0 and <10.0 ng/mL must have documentation of a negative histologic biopsy of carcinoma of the prostate within 12 months prior to screening.

Exclusion Criteria:

* History of radical prostatectomy, or other pelvic surgery or procedure, including any pelvic surgical procedure on the urinary tract apart from transurethral resection, pelvic surgery for malignancy or bowel resection, or a history of lower urinary tract malignancy or trauma. History of urinary retention or lower urinary tract (bladder) stones within 6 months of screening.
* Current or previous history of malignant disease of the prostate.
* Concomitant treatment with or ingestion of cytochrome P 450 3A4 (CYP3A4)-inducing or -inhibiting agents from 2 weeks prior to dosing and through the end of the study. Including herbal/food and other supplements, fruit, or fruit juices containing grapefruit or pomegranate components.
* History of loss of vision in one eye because of nonarteritic anterior ischemic optic neuropathy (NAION), regardless of whether this episode was in connection or not with previous PDE5 inhibitor exposure.
* Subjects with chronic stable angina treated with long-acting nitrates, subjects with chronic stable angina who required short-acting nitrates in the 90 days prior to screening visit, or subjects with angina occurring during sexual intercourse in the 6 months prior to screening.
* Subjects having met the criteria for unstable angina within 6 months prior to screening, history of myocardial infarction or coronary artery bypass graft surgery within 90 days prior to screening, or percutaneous coronary intervention (for example, angioplasty or stent placement) within 90 days prior to screening.
* Any evidence of heart disease (New York Heart Association [NYHA] greater than or equal to Class III) within 6 months of screening.
* A history of cardiac arrest.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-07; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Munich, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Japanese Participants: Japanese participants who received 5 mg of tadalafil once daily for 10 days
- Caucasian Participants: Caucasian participants who received 5 mg of tadalafil once daily for 10 days
Period: Overall Study
Arm/Group | Japanese Participants | Caucasian Participants
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Japanese Participants | Caucasian Participants | Total
Number analyzed (Participants) | 12 | 12 | 24
Age Continuous [Mean (Standard Deviation); unit: years] | 57.0 (9.9) | 60.6 (7.2) | 58.8 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 12 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 12 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 12 | 0 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 12 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 0 | 12 | 12
  Japan | 12 | 0 | 12

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Area Under the Concentration Curve (AUC) for Tadalafil and Metabolite IC710
Description: AUC for Day 1 is reported as AUC(tau [t], day 1), which is AUC from time zero to 24 hours (t) postdose on Day 1. AUC for Day 10 is reported as AUC(t,steady state [ss]), which is AUC during one 24-hour dosing interval at steady-state.
Time Frame: 1 day and 10 days
Population: All enrolled participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter (ng*hr/mL)
Arm/Group | Japanese Participants | Caucasian Participants
Number analyzed (Participants) | 12 | 12
nanograms*hour/milliliter (ng*hr/mL)
  Day 1 Tadalafil | 1410 (31) | 1340 (17)
  Day 10 Tadalafil | 2710 (27) | 3410 (51)
  Day 1 Metabolite IC710 | 525 (27) | 399 (23)
  Day 10 Metabolite IC710 | 2270 (30) | 2290 (48)
Statistical Analysis 1: Comparison: Japanese Participants vs Caucasian Participants; Test type: Superiority or Other; Ratio of Geometric Least Squares Means = 1.05, 90% CI 2-sided [0.84 to 1.32] — Day 1 Tadalafil Ratio of Geometric Least Squares Means (Japanese/Caucasian)
Statistical Analysis 2: Comparison: Japanese Participants vs Caucasian Participants; Test type: Superiority or Other; Ratio of Geometric Least Squares Means = 0.80, 90% CI 2-sided [0.64 to 1.00] — Day 10 Tadalafil Ratio of Geometric Least Squares Means (Japanese/Caucasian)
Statistical Analysis 3: Comparison: Japanese Participants vs Caucasian Participants; Test type: Superiority or Other; Ratio of Geometric Least Squares Means = 1.31, 90% CI 2-sided [1.05 to 1.64] — Day 1 Metabolite IC710 Ratio of Geometric Least Squares Means (Japanese/Caucasian)
Statistical Analysis 4: Comparison: Japanese Participants vs Caucasian Participants; Test type: Superiority or Other; Ratio of Geometric Least Squares Means = 0.99, 90% CI 2-sided [0.79 to 1.24] — Day 10 Metabolite IC710 Ratio of Geometric Least Squares Means (Japanese/Caucasian)

2. Primary Outcome: Pharmacokinetics: Concentration Maximum (Cmax) of Tadalafil and Metabolite IC710
Time Frame: 1 day and 10 days
Population: All enrolled participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Japanese Participants | Caucasian Participants
Number analyzed (Participants) | 12 | 12
nanograms per milliliter (ng/mL)
  Day 1 Tadalafil | 102 (27) | 104 (19)
  Day 10 Tadalafil | 173 (24) | 215 (36)
  Day 1 Metabolite IC710 | 32.1 (25) | 24.0 (26)
  Day 10 Metabolite IC710 | 105 (31) | 102 (47)
Statistical Analysis 1: Comparison: Japanese Participants vs Caucasian Participants; Test type: Superiority or Other; Ratio of Geometric Least Squares Means = 0.98, 90% CI 2-sided [0.81 to 1.18] — Day 1 Tadalafil Ratio of Geometric Least Squares Means(Japanese/Caucasian)
Statistical Analysis 2: Comparison: Japanese Participants vs Caucasian Participants; Test type: Superiority or Other; Ratio of Geometric Least Squares Means = 0.81, 90% CI 2-sided [0.67 to 0.97] — Day 10 Tadalafil Ratio of Geometric Least Squares Means (Japanese/Caucasian)
Statistical Analysis 3: Comparison: Japanese Participants vs Caucasian Participants; Test type: Superiority or Other; Ratio of Geometric Least Squares Mean = 1.33, 90% CI 2-sided [1.07 to 1.67] — Day 1 Metabolite IC710 Ratio of Geometric Least Squares Means (Japanese/Caucasian)
Statistical Analysis 4: Comparison: Japanese Participants vs Caucasian Participants; Test type: Superiority or Other; Ratio of Geometric Least Squares Means = 1.03, 90% CI 2-sided [0.83 to 1.29] — Day 10 Metabolite IC710 Ratio of Geometric Least Squares Means (Japanese/Caucasian)

3. Primary Outcome: Pharmacokinetics: Time to Concentration Maximum (Tmax) of Tadalafil and Metabolite IC710
Time Frame: 1 day and 10 days
Population: All enrolled participants
Measure: Median (Full Range); unit: hours
Arm/Group | Japanese Participants | Caucasian Participants
Number analyzed (Participants) | 12 | 12
hours
  Day 1 Tadalafil | 4.00 [1.00 to 4.00] | 2.00 [1.00 to 4.00]
  Day 10 Tadalafil | 3.00 [2.00 to 4.00] | 2.53 [1.00 to 4.00]
  Day 1 Metabolite IC710 | 23.83 [23.83 to 23.83] | 24.00 [16.02 to 24.03]
  Day 10 Metabolite IC710 | 4.00 [0.00 to 24.00] | 8.00 [0.00 to 24.00]
Statistical Analysis 1: Comparison: Japanese Participants; Test type: Superiority or Other; Wilcoxon (Mann-Whitney); Tadalafil Median Difference (Day 1 - Day 10) in Japanese Participants; Median Difference (Final Values) = 0.00
Statistical Analysis 2: Comparison: Caucasian Participants; Test type: Superiority or Other; Wilcoxon (Mann-Whitney); Tadalafil Median Difference (Day 1 - Day 10) in Caucasian Participants; Median Difference (Final Values) = 0.00
Statistical Analysis 3: Comparison: Japanese Participants; Test type: Superiority or Other; Wilcoxon (Mann-Whitney); Metabolite IC710 Median Difference (Day 1 - Day 10) in Japanese participants; Median Difference (Final Values) = 19.83
Statistical Analysis 4: Comparison: Caucasian Participants; Test type: Superiority or Other; Wilcoxon (Mann-Whitney); Metabolite IC710 Median Difference (Day 1 - Day 10) in Caucasian participants; Mean Difference (Final Values) = 16.02

ADVERSE EVENTS:
Arm/Group | Japanese Participants | Caucasian Participants
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 12/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Japanese Participants (N=12) | Caucasian Participants (N=12)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2)
Bowel movement irregularity (Gastrointestinal disorders) | 0 (0) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (4)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2)
Chest pain (General disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 4 (4)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days